CLINICAL TRIAL: NCT00450671
Title: Seton Placement vs. Surgisis Anal Fistula Plug Insertion for Perirectal Fistula: A Prospective Randomized Study
Brief Title: Treatment of Perirectal Fistula With Cutting Seton vs. Collagen Plug
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Seton vs. Surgisis; HS-06-00342 (Other: USC IRB)
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Anal Fistula
Keywords: Fistula-in-ano; Anal fistula; Perirectal fistula; Collagen plug; Surgisis; Seton
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Collagen Plug Placement
Procedure: Seton placement

SUMMARY:
The purpose of this study is to determine if the collagen plug method heals perirectal fistulae as well as the conventional seton method.

DETAILED DESCRIPTION:
Traditional treatments for transsphincteric perirectal fistulae rely upon an immediate (fistulotomy) or delayed (seton) transsection of the sphincter muscle possibly resulting in fecal incontinence, take a long time to heal, and/or are associated with significant failure rates (ex. fibrin glue).

Newer treatment concepts such as the collagen plug do not physically interrupt the sphincter muscle, avoid and minimize the risk of fecal incontinence, and decrease the time to fistula healing. Exciting initial reports have confirmed the collagen plug's utility in treating perirectal fistulae, but a systematic scientific comparison is needed to validate the new, less invasive plug method.

The primary goal of this study is to show that the collagen plug heals transsphincteric perirectal fistulae as well as the conventional seton method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that are undergoing surgery for perirectal fistulae by the USC Colorectal Group
2. Patients that are older than 18 years of age and are able to understand and sign consent
3. Patients that are suitable candidates for either seton or collagen plug placement

Exclusion Criteria:

1. Preoperative patient exclusion factors:

   * Pregnant patients
   * Patients with a tumor-related fistula
   * Patients with known allergies to porcine products
   * Patients with known Crohn's disease
2. Intraoperative patient exclusion factors:

   * Patients with an active purulent infection (pus draining from the fistula tract or abscess associated with the fistula tract) at the time of surgery
   * Patients with a large diameter fistula (>3mm)
   * Patients with a superficial fistula
   * Patients with a short fistula (<1 cm in length)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-02; Study Completion 2013-05-09 (Actual)

PRIMARY OUTCOMES:
Fistula healing
Treatment failure

SECONDARY OUTCOMES:
Time to fistula healing
Time to treatment failure
Rates of postoperative fecal continence

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Kaiser, MD, Principal Investigator — University of Southern California Department of Colorectal Surgery
Locations (4):
- United States (4):
  - H.Claude Hudson Comprehensive Health Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC Norris Cancer Center, Los Angeles, California
  - USC/University Hospital, Los Angeles, California

REFERENCES:
- [Background] Zmora O, Neufeld D, Ziv Y, Tulchinsky H, Scott D, Khaikin M, Stepansky A, Rabau M, Koller M. Prospective, multicenter evaluation of highly concentrated fibrin glue in the treatment of complex cryptogenic perianal fistulas. Dis Colon Rectum. 2005 Dec;48(12):2167-72. doi: 10.1007/s10350-005-0199-1. PMID 16258708
- [Background] Champagne BJ, O'Connor LM, Ferguson M, Orangio GR, Schertzer ME, Armstrong DN. Efficacy of anal fistula plug in closure of cryptoglandular fistulas: long-term follow-up. Dis Colon Rectum. 2006 Dec;49(12):1817-21. doi: 10.1007/s10350-006-0755-3. PMID 17082891
- [Background] Johnson EK, Gaw JU, Armstrong DN. Efficacy of anal fistula plug vs. fibrin glue in closure of anorectal fistulas. Dis Colon Rectum. 2006 Mar;49(3):371-6. doi: 10.1007/s10350-005-0288-1. PMID 16421664